CLINICAL TRIAL: NCT00646178
Title: Multicenter Study of the Safety and Efficacy of the Human Anti-TNF Monoclonal Antibody Adalimumab in Subjects With Moderate to Severely Active Psoriatic Arthritis Subjects With Inadequate Response to Disease Modifying Anti-Rheumatic Drug Therapy
Brief Title: Study of the Safety and Efficacy of Adalimumab in Subjects With Moderate to Severely Active Psoriatic Arthritis Subjects With Inadequate Response to Disease Modifying Anti-Rheumatic Drug Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Beverly Paperiello / Director, Clinical Research Development, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-570
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Arthritis; Psoriatic
MeSH Terms: conditions — Arthritis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: adalimumab
- B (Placebo Comparator)
  Interventions: Drug: placebo for adalimumab

INTERVENTIONS:
Drug: adalimumab — 40 mg adalimumab eow Week 0 - Week 12
  Other Names: ABT-D2E7; Humira
  Arms: A
Drug: placebo for adalimumab — placebo eow Week 0 - Week 12
  Other Names: placebo
  Arms: B

SUMMARY:
Multicenter Study of the Safety and Efficacy of Adalimumab in Subjects with Moderate to Severely Active Psoriatic Arthritis Subjects with Inadequate Response to Disease Modifying anti-Rheumatic Drug Therapy

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe PsA
* Inadequate response to DMARD therapy
* Corticosteroid stable dose <=10 mg QD
* DMARDs must have been taken for 3 months and stable dose for 4 weeks
* MTX maximum dose = <=30 mg/week
* Active chronic plaque PS or documented history of chronic plaque PS

Exclusion Criteria:

* No other active skin disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-06; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
ACR20 | Week 12
Adverse Events | Throughout the Study

SECONDARY OUTCOMES:
ACR50/70 | Week 12
Modified Psoriatic Arthritis Response Criteria | Week 12
Multiple QOL Assessments | Week 12
Physicians Global Assessment for Psoriasis | Week 12